CLINICAL TRIAL: NCT03245099
Title: Management of Non Convulsive Status Epilepticus
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rewaa Mohammed, Principlal investigator, Assiut University
Other Study IDs: MONCSE
Record Dates: First submitted 2017-08-04; First posted 2017-08-10 (Actual); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Status Epilepticus
MeSH Terms: conditions — Status Epilepticus | interventions — Cross-Sectional Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: cross sectional — Electroencephalograph will be done to all patients who fulfill the inclusion criteria to detect presence of electrical discharge with in the brain.Complete blood count ,liver function test ,kidney function test ,blood glucose level and serum electrolytes will be done to selected cases according to the clinical presentation

SUMMARY:
Non convulsive status epilepticus is a persistent change in behavioural and or mental process from baseline associated with continuous epileptiform activity in electroencephalograph,it occur in about 50 percent in patients with coma and convulsions and in 8-13 percent in intensive care unit patients

DETAILED DESCRIPTION:
Early recognition and treatment of non convulsive status epilepticus are essential to optimize response to treatment and to prevent neurological sequelae, over diagnosis and aggressive use of anticonvulsants can contribute to morbidity and mortality.It displays great diversity in response to anticonvulsants,therefore treatment in intensive care units is required for selected cases .The aetiology and clinical forms are strong predictors for the overall prognosis.Treatment is poorly understood and follows the standard regimen for convulsive status epilepticus

ELIGIBILITY:
Inclusion Criteria:

* patients who have generalized tonic colonic convulsions and prolonged post ictal state more than 30 minutes
* patients presented with un explained psychic or speech disorder
* patients presented with stupor or confusion
* Patients presented with un explained coma

Exclusion Criteria:

* patients with progressive neurological disease
* Patients with severe cerebral anoxia
* Patients with liver or hepatic impairment

Ages: 12 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: * Patients 1-18 years
  * Generalized tonic clonic convulsions and prolonged post ictal period more than 30 minutes
  * Un explained coma ,stupor,confusion and psychic or speech disorder
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-12 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Number of cured patients | An average of 1 year
  Number of cured patients

CONTACTS AND LOCATIONS:
Overall Officials: Rewaa Mohammed, MD, Principal Investigator — Assiut University
Locations (1):
- AssiutU, Asyut, Egypt